CLINICAL TRIAL: NCT05924698
Title: Effects of Blood Flow Restriction Therapy Combined With Neuromuscular Electrostimulation in Amateur Female Soccer Players: A Pilot Study
Brief Title: Blood Flow Restriction Therapy Combined With Neuromuscular Electrostimulation in Amateur Female Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Extremadura (Other)
Responsible Party: Principal Investigator, Carlos Fernández-Morales, Clinical Professor, Universidad de Extremadura
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04
Record Dates: First submitted 2023-06-13; First posted 2023-06-29 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Knee
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation; Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): This arm only received the Neuromuscular and Muscular Electrical Stimulation (NMES) intervention.
  Interventions: Other: Electrostimulation
- Experimental group (Experimental): This arm received the intervention with NMES and Blood flow restriction (BFR).
  Interventions: Other: Electrostimulation; Other: Blood flow restriction therapy

INTERVENTIONS:
Other: Electrostimulation — Consisting of the use of NMES (biphasic symmetrical pulse, bipolar mode, 50Hz frequency, pulse duration 300 μs at 1:1 ratio) (S82®; Enraf-Nonius BV, Rotterdam, The Netherlands). The self-adhesive electrodes (8x5 cm2 Pals Platinum © type, Axelgaard Manufacturing Co. Ltd, Fallbrook, CA, USA) were placed on the quadriceps muscle. The positives electrodes placed distally on the rectus anterior and vastus externus and negative electrodes were placed proximally on the rectus anterior and vastus internus. The over current program consisted of 8 seconds (s) of work (ON phase) and 8 seconds of rest (OFF phase). The overcurrent program in the ON phase had a rise time of 2 s, a hold time of 4 s and a fall time of 2 s. The intensity of the electric current was increased to the maximum perceived tolerance, achieving a clear contraction without producing fatigue.
Other: Blood flow restriction therapy — To attain partial vascular occlusion, a PTS ii portable tourniquet system (Delphi Medical, Vancouver, BC, Canada) with a corresponding size-specific tourniquet was placed around the patient's proximal thigh. This system allows for precise control of cuff pressure throughout training despite the changes in muscle volume that naturally occur while performing exercises. Total limb occlusion pressure (LOP) was identified by determining the pressure required to eliminate a detectable pulse using Doppler ultrasound. Partial vascular occlusion was achieved by setting the tourniquet to 80% of the LOP. This ensured that venous occlusion was obtained while still allowing arterial inflow and was personalized to each patient despite variations in thigh girth, cuff size, and systolic blood pressure. An Easy-Fit Tourniquet Cuff (Delfi Medical, Vancouver, VC, Canada) was used with the PTS ii system.
  Arms: Experimental group

SUMMARY:
The objective is to know the effects of Neuromuscular Electrical Stimulation (NMES) and its combination with Blood Flow Restriction (BFR) Therapy in healthy amateur female soccer players.

DETAILED DESCRIPTION:
The objective is to know the effects of Neuromuscular Electrical Stimulation (NMES) and its combination with Blood Flow Restriction (BFR) Therapy in healthy amateur female soccer players.

For this purpose, a randomized clinical trial will be performed: 20 amateur female soccer players were distributed in two groups (control group n=10; experimental group n=10). In the control group, NMES (symmetrical biphasic rectangular pulse, 350 μs and 80Hz) combined simultaneously with active exercise in knee extension (75 repetitions in 4 sets, 20% 1RM, 30 seconds rest between sets) was applied. The experimental group performed the same intervention combined with blood flow restriction (BFR) therapy (80% of arterial occlusion pressure). The variables measured were muscle strength, muscle volume and static proprioception.

ELIGIBILITY:
Inclusion Criteria:

* Be federated in a sports club playing 11-a-side soccer for at least the last two seasons.
* Be between 16 and 28 years of age.
* Be physically active players at the time of the study with a regular practice of at least 5 hours per week during the last 2 months,
* Have been playing soccer for at least 5 hours per week during the last 2 months.
* Have been playing soccer for at least 2 years

Exclusion Criteria:

* Those who presented at the time of the study any lesion classified according to the Munich consensus and diagnosed by a doctor.
* Those with systemic lupus erythematosus.
* Hemophilia.
* Unregulated hypertension.
* History of pulmonary thromboembolism or stroke.
* Impaired blood coagulation.
* Contraceptive intake.
* Spinal radicular lesions.
* Previous surgeries related to the circulatory system.

Ages: 16 Years to 28 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Amateur 11-a-side soccer players
Enrollment: 20 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-06-13 (Actual)

PRIMARY OUTCOMES:
Muscular Strenght | During the intervention, at day 1
  It was performed using an isokinetic dynamometer (Kineo, Globus, Codognè, Italy). The maximum peak force that the user can perform was measured by means of the concentric-eccentric isokinetic force test. The patient is placed seated on the seat of the machine and with the dominant lower limb, performs 5 contractions with the maximum force, obtaining the concentric and eccentric peak force.
Muscle volume | During the intervention, at day 1
  It was performed by means of the thigh perimeter, using a tape measure. The superior pole of the patella is selected as an anatomical reference point and four segments are marked from it, located at 5, 10, 15 and 20 centimeters respectively (95). Subsequently, placing the beginning of the measuring tape at the mark of the segment in question, the thigh is encircled keeping the beginning of the tape fixed, which will coincide with a measurement of the tape when it is reached. This measurement is taken before the start of the quadriceps work with the knee extension exercise and at the end of the 15 minutes of rest after this work.

SECONDARY OUTCOMES:
Knee joint repositioning | During the intervention, at day 1
  It was performed through the ability to perceive and reproduce an articular angle previously represented and explained passively. The angles are photographed and measured using the SAPO® computer program, by means of the placement of four marked points on the greater trochanter, lateral epicondyle of the femur, head of the fibula and peroneal malleolus. To perform this procedure, the user must memorize two positions, knee flexion of 90º and knee flexion of 135º, taking 3 photographs of each position in both seated and prone positions.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Espejo-Antúnez, Ph.D., Study Director — University of Extremadura
Locations (1):
- University of Extremadura, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: No